CLINICAL TRIAL: NCT02114151
Title: A Phase 3, Multicenter, Open-Label, Single-Arm Study to Investigate the Efficacy and Safety of a 12-Week Regimen of Simeprevir in Combination With Sofosbuvir in Treatment-Naïve or -Experienced Subjects With Chronic Genotype 1 Hepatitis C Virus Infection and Cirrhosis
Brief Title: Efficacy and Safety Study of Simeprevir in Combination With Sofosbuvir in Participants With Genotype 1 Chronic Hepatitis C Virus Infection and Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR103431; TMC435HPC3018 (Other: Janssen Infectious Diseases BVBA)
Record Dates: First submitted 2014-04-02; First posted 2014-04-15 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C Virus Infection; Simeprevir; Sofosbuvir; HCV; Cirrhosis
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Simeprevir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Simeprevir/Sofosbuvir) (Experimental): 100 participants will receive 1 capsule of 150 mg simeprevir and 1 tablet of 400 mg sofosbuvir orally (by mouth) once daily for 12 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Simeprevir — 100 participants will receive 1 capsule of 150 mg orally once daily for 12 weeks.
Drug: Sofosbuvir — 100 participants will receive 1 tablet of 400 mg sofosbuvir orally once daily for 12 weeks.

SUMMARY:
The purpose of the study is to investigate the efficacy and safety of 12 weeks of simeprevir (150 mg qd) in combination with sofosbuvir (400 mg qd) in chronic hepatitis C virus (HCV) genotype 1 infected men and women with cirrhosis who are HCV treatment-naïve or treatment-experienced.

DETAILED DESCRIPTION:
This is a open-label (all people know the identity of the intervention), single arm, multicenter study. The study will consist of a screening phase up to 4 weeks, open-label treatment phase of 12 weeks, and post-treatment follow up phase up to 24 weeks after end of treatment. Approximately 100 participants will receive 150 mg simeprevir in combination with 400 mg sofosbuvir once dailyfor 12 weeks. Safety evaluations will include assessment of adverse events, clinical laboratory tests, vital signs, and physical examination. The maximum study duration for each participant will be approximately 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus (HCV) genotype 1 infection (confirmed at screening).
* HCV ribonucleic acid (RNA) greater than 10,000 IU/mL at screening
* Treatment-experienced participants must have at least 1 documented previous course of interferon-based regimen with or without ribavirin
* Participants must have an hepatic imaging procedure (ultrasound, computerized tomography scan or magnetic resonance imaging scan) within 6 months prior to the screening visit (or between screening and Day 1) with no findings suspicious for hepatocellular carcinoma
* Participant must be willing and able to comply with the protocol requirements
* Participants with liver cirrhosis

Exclusion Criteria:

* Evidence of clinical hepatic decompensation (history or current evidence of ascites, bleeding varices or hepatic encephalopathy)
* Infection/co-infection with HCV non-genotype 1
* Co-infection with human immunodeficiency virus (HIV) type 1 or type 2 (HIV-1 or HIV-2) (positive HIV-1 or HIV-2 antibodies test at screening)
* Co-infection with hepatitis B virus (hepatitis B-surface-antigen positive)
* Previously been treated with any direct acting anti-HCV agent (approved or investigational) for chronic HCV infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (34):
- United States (32):
  - Dothan, Alabama
  - Bakersfield, California
  - Chula Vista, California
  - Los Angeles, California
  - San Diego, California
  - Englewood, Colorado
  - Bradenton, Florida
  - Lauderdale Lakes, Florida
  - Maitland, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Marietta, Georgia
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Hillsborough, New Jersey
  - Vineland, New Jersey
  - New York, New York
  - Asheville, North Carolina
  - Winston-Salem, North Carolina
  - East Greenwich, Rhode Island
  - Providence, Rhode Island
  - Greer, South Carolina
  - Germantown, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
- Canada (2):
  - Vancouver, British Columbia
  - Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 147 participants from the United States and Canada were Screened and 103 were enrolled into the study. All 103 participants who received at least 1 dose of study drug and so were included in intent to treat (ITT) population.
Groups:
- Simeprevir Plus Sofosbuvir: Participants received simeprevir 150 milligram (mg) in combination with sofosbuvir 400 mg once daily for 12 weeks.
Period: Overall Study
Arm/Group | Simeprevir Plus Sofosbuvir
Started | 103
Completed | 96
Not Completed | 7
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 103
Age, Continuous [Median (Full Range); unit: years] | 58 [29 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Sustained Virologic Response (SVR) 12 Weeks After the Actual End of Treatment (EOT)
Description: Participants with hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) 25 international unit per milliliter (IU/mL) (detectable or undetectable) at 12 weeks after the actual end of treatment.
Time Frame: Week 24
Population: Intent-to-treat (ITT) population included all enrolled participants who took at least 1 dose of investigational medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 103
Percentage of Participants | 83.5 [75.8 to 91.1]

2. Secondary Outcome: Percentage of Participants With a Sustained Virologic Response (SVR) 4 Weeks After the Actual End of Treatment (EOT)
Description: Participants with hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) 25 international unit per milliliter (IU/mL) (detectable or undetectable) at 4 weeks after the actual end of treatment.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 103
Percentage of Participants | 86.4 [79.3 to 93.5]

3. Secondary Outcome: Percentage of Participants With a Sustained Virologic Response (SVR) 24 Weeks After the Actual End of Treatment (EOT)
Description: Participants with hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) 25 international unit per milliliter (IU/mL) (detectable or undetectable) at 24 weeks after the actual end of treatment.
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 103
Percentage of Participants | 82.5 [74.7 to 90.3]

4. Secondary Outcome: Percentage of Participants With On-treatment Virologic Response
Description: On-treatment virologic response was determined by HCV RNA results satisfying a specified threshold. <LLOQ undetectable was considered as threshold at any time point. The LLOQ value is 25 IU/mL. EOT=End of Treatment.
Time Frame: Week 2, 4 and End of Treatment (Week 12)
Population: Intent-to-treat (ITT) population included all enrolled participants who took at least 1 dose of investigational medication. Here 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Number; unit: Percentage of Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 103
Percentage of Participants
  Week 2: < 100 IU/mL (n=102) | 90.2
  Week 2: < 25 IU/mL (n=102) | 68.6
  Week 2: < 25 IU/mL Detectable (n=102) | 44.1
  Week 2: < 25 IU/mL Undetectable (n=102) | 24.5
  Week 4: < 100 IU/mL (n=102) | 99.0
  Week 4: < 25 IU/mL (n=102) | 99.0
  Week 4: < 25 IU/mL Detectable (n=102) | 15.7
  Week 4: < 25 IU/mL Undetectable (n=102) | 83.3
  EOT (Week 12): < 100 IU/mL (n=103) | 97.1
  EOT (Week 12): < 25 IU/mL (n=103) | 97.1
  EOT (Week 12): < 25 IU/mL Detectable (n=103) | 0
  EOT (Week 12): < 25 IU/mL Undetectable (n=103) | 97.1

5. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: On-treatment failure is defined as participants who do not achieve SVR12 and with confirmed detectable HCV RNA at the actual end of study drug treatment.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all randomized participants who took at least one dose of investigational drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 103
Percentage of Participants | 2.9

6. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as confirmed greater than (>) 1 log10 increase in HCV RNA from nadir or confirmed HCV RNA >100 IU/mL in participants who had previously achieved HCV RNA < LLOQ (25 IU/mL).
Time Frame: Up to End of Treatment (Week 12)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 103
Percentage of Participants | 1.9

7. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as participants who did not achieve SVR12 and had HCV RNA < LLOQ (25 IU/mL) undetectable at EOT and had HCV RNA >= LLOQ (25 IU/mL) during the follow-up period.
Time Frame: During the Follow-up (Week 24)
Population: Intent-to-treat (ITT) population included all enrolled participants who took at least 1 dose of investigational medication. Here "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 99
Percentage of Participants | 13.1

8. Secondary Outcome: Change From Baseline in Hepatitis C Symptom and Impact Questionnaire Version 4 (HCV-SIQv4) Overall Body System Score (OBSS) up to Follow-up Week 12
Description: The HCV-SIQv4 OBSS was a self-administered questionnaire that contained 33 items: 29 questions developed to assess severity or frequency of symptoms associated with HCV or its treatment, 3 questions regarding the impact of symptoms on work/school attendance, and 1 question regarding the impact of symptoms on daily activities. A symptom severity score (the mean of responses to the 29 symptom items); each symptom score was transformed to have a range from 0 to 100 (most severe). Higher HCV SIQv4 scores indicates worse symptom severity, more time missed from work/school, and more impairment in daily activities, respectively.
Time Frame: Baseline, Week 4, Week 12 and Follow-Up Week 12
Population: Intent-to-treat (ITT) population included all enrolled participants who took at least 1 dose of investigational medication. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure and 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 98
Units on a Scale
  Baseline (n=98) | 17.4 (1.47)
  Change at Week 4 (n=96) | -4.9 (1.23)
  Change at Week 12 (n=89) | -4.7 (1.39)
  Change at Follow-up Week 12 (n=94) | -5.8 (1.36)

9. Secondary Outcome: Change From Baseline in Fatigue Severity Score (FSS) up to Follow-up Week 24
Description: The FSS was a self-administered questionnaire with 9 items developed to assess disabling fatigue that has been used extensively in studies of chronic HCV infection. Item responses were measured on a 7-point Likert scale ranging from strongly disagree (1 point) to strongly agree (7 points). The 9 items were averaged to produce a total score; a lower total score indicates less severe fatigue. FSS scores have a range from 1 to 7 where higher scores indicate more severe fatigue.
Time Frame: Baseline, Week 12, Follow-up Week 12 and 24
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 96
Units on a Scale
  Baseline (n=96) | 3.4 (0.18)
  Change at Week 12 (n=86) | -0.4 (0.18)
  Change at Follow-up Week 12 (n=92) | -0.6 (0.16)
  Change at Follow-up Week 24 (n=86) | -0.8 (0.18)

10. Secondary Outcome: Percentage of Participants With Depression by Using Center for Epidemiologic Studies Depression Scale (CES-D)
Description: The CES-D Scale assessed how often during the past week participants experienced 20 symptoms commonly associated with major depression. The CES-D scores range from 0 (no symptoms) to 60 (all 20 symptoms most or all of the time during the past 5 to 7 days). The CES-D scores between 16 and 23 points indicate mild to moderate depressive illness while CES-D scores >=23 indicate probable major depressive illness.
Time Frame: Baseline, Week 12, Follow-up Week 12 and 24
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 96
Percentage of Participants
  Baseline: No Depression (n=96) | 67.7
  Baseline: Mild to Moderate Depression (n=96) | 16.7
  Baseline: Severe Depression (n=96) | 15.6
  Week 12: No Depression (n=88) | 77.3
  Week 12: Mild to Moderate Depression (n=88) | 15.9
  Week 12: Severe Depression (n=88) | 6.8
  Follow-up Week 12: No Depression (n=94) | 79.8
  Follow-up Week12:Mild to Moderate Depression(n=94) | 6.4
  Follow-up Week 12: Severe Depression (n=94) | 13.8
  Follow-up Week 24: No Depression (n=88) | 79.5
  Follow-up Week24:Mild to Moderate Depression(n=88) | 10.2
  Follow-up Week 24: Severe Depression (n=88) | 10.2

11. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension Questionnaire (EQ-5D) up to Follow-up Week 24
Description: The EQ-5D questionnaire was a brief, generic health-related quality of life (HRQOL) assessment that could also be used to incorporate participant preferences into health economic evaluations. The EQ-5D questionnaire assessed HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a "thermometer" visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Time Frame: Baseline, Follow-up Week 12 and 24
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 96
Units on a Scale
  Baseline (n=96) | 70.1 (2.17)
  Change at Follow-up Week 12 (n=92) | 9.8 (1.90)
  Change at Follow-up Week 24 (n=86) | 9.5 (1.75)

12. Secondary Outcome: Number of Participants Not Achieving SVR Showing Emerging Mutation at Time of Failure in HCV NS3/4A Sequence and NS5B up to Follow-up Week 24
Description: Sequencing of the HCV nonstructural protein 3/4A (NS3/4A) and nonstructural protein 5B (NS5B) genes was done to identify pre-existing sequence polymorphisms and characterize emerging HCV viral variants in participants not achieving SVR. Sequencing data is available for 16 participants.
Time Frame: Baseline, Day 3, Week 1, 2, 3, 4, 8, 12, Follow-up Week 4, 12 and 24
Population: Intent-to-treat (ITT) population included all enrolled participants who took at least 1 dose of investigational medication. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Simeprevir Plus Sofosbuvir
Number analyzed (Participants) | 16
Participants
  HCV NS3 | 13
  NS5B | 0

ADVERSE EVENTS:
Time Frame: Baseline up to End of Treatment (Week 36)
Arm/Group | Simeprevir Plus Sofosbuvir
Serious Adverse Events (participants affected / at risk) | 5/103
Other Adverse Events (participants affected / at risk) | 47/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simeprevir Plus Sofosbuvir (N=103)
Cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Non-cardiac chest pain (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simeprevir Plus Sofosbuvir (N=103)
Fatigue (General disorders) | 21
Headache (Nervous system disorders) | 21
Nausea (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 8
Insomnia (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.